CLINICAL TRIAL: NCT07366580
Title: TOUCHMinds: An RCT on Help-seeking for Adolescent Anxiety
Brief Title: TOUCHminds: Help-seeking in Adolescents With Anxiety
Acronym: TOUCHminds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: Foundation for Science and Technology (Unknown)
Responsible Party: Principal Investigator, Paula Vagos, PhD, Aveiro University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2024.05050.BD; 2024.05050.BD (Other Grant/Funding Number: Foundation for Science and Technology, Portugal)
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Anxiety Symptoms; Anxiety Disorders
Keywords: Anxiety; Adolescents; Help-seeking; Web-based intervention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This investigation comprises two sequential studies. Study I (feasibility) is a single-arm, pre-post study design with two intervention groups (clinical, n=5; subclinical, n=5), both receiving the TOUCHminds. Study I will assess recruitment procedures, dropout rates, usage patterns, therapist fidelity, acceptability, usability, satisfaction, and preliminary effects. Study II (RCT) is a randomized, controlled, parallel-group trial evaluating the effectiveness of the TOUCHminds in adolescents with clinical and subclinical anxiety symptoms. Participants will be randomly assigned to one of four conditions: Clinical Intervention (n = 24), Clinical Control (n = 24), Subclinical Intervention (n = 24), or Subclinical Control (n = 24).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Clinical Group (study I and study II) (Experimental): Adolescents meeting diagnostic criteria for one or more anxiety disorders (study I n= 5; study II n = 24). Participants receive the TOUCHminds intervention. Assessments are conducted at pre-intervention (study I and II), post-intervention (9 weeks later; study I and II), and at 3-month follow-up (study II).
  Interventions: Behavioral: TOUCHminds - Web-Based Intervention
- Control: Clinical Group (study II) (No Intervention): Adolescents meeting diagnostic criteria for one or more anxiety disorders (study II n = 24). Participants do not receive the intervention during the main study period but are assessed at the same time points as the intervention group: pre-intervention, post-intervention (9 weeks later), and 3-month follow-up. After completing the final assessment, they are granted access to the TOUCHminds intervention.
- Experimental: Subclinical Group (study I and study II) (Experimental): Adolescents presenting subclinical anxiety symptoms (i.e., high self-reported anxiety but no mental disorder diagnosis; study I n= 5; study II n = 24). Participants receive the TOUCHminds intervention. Assessments are conducted at pre-intervention (study I and II), post-intervention (9 weeks later; study I and II), and at 3-month follow-up (study II).
  Interventions: Behavioral: TOUCHminds - Web-Based Intervention
- Control: Subclinical Group (study II) (No Intervention): Adolescents presenting subclinical anxiety symptoms (i.e., high self-reported anxiety but no mental disorder diagnosis; study II n = 24). Participants do not receive the intervention during the main study period but are assessed at the same time points as the intervention group: baseline (pre-intervention), post-intervention (9 weeks later), and 3-month follow-up. After completing the final assessment, they are granted access to the TOUCHminds intervention.

INTERVENTIONS:
Behavioral: TOUCHminds - Web-Based Intervention — A web-based intervention designed to promote help-seeking in adolescents with clinical or subclinical anxiety symptoms. The program combines six self-guided online modules with three individual videoconference sessions with a trained psychologist. It integrates core components from Cognitive Behavioral Therapy (CBT), Acceptance and Commitment Therapy (ACT), Compassion-Focused Therapy (CFT), Motivational Interviewing, and the Transtheoretical Model of Change. The intervention is tailored to the developmental stage of adolescents and is delivered remotely to participants meeting the inclusion criteria.
  Arms: Experimental: Clinical Group (study I and study II); Experimental: Subclinical Group (study I and study II)

SUMMARY:
Adolescents frequently experience clinical and subclinical anxiety symptoms, yet many avoid seeking professional help. While universal interventions exist to promote help-seeking, targeted programs for adolescents with elevated anxiety symptoms remain scarce. Therefore, accessible and tailored strategies are needed to effectively promote help-seeking among this group.

TOUCHminds is a web-based intervention designed to enhance help-seeking among adolescents with clinical or subclinical anxiety. The program consists of six self-guided modules featuring interactive activities (e.g., images, videos, simulation activities, and audio recordings), combined with three synchronous sessions led by a psychologist via videoconference. The intervention explicitly targets precursors of help-seeking, including mental health literacy, mental health stigma, self-compassion, readiness to change, and stage of change.

This research project comprises two studies. Study I, a feasibility study involving 10 adolescents aged 15 to 17, will assess recruitment procedures, dropout rates, usage patterns, therapist fidelity, acceptability, usability, satisfaction, and preliminary effects. Study II, a randomized controlled trial (RCT), intends to include 96 adolescents randomly assigned to four groups: clinical intervention, clinical control, subclinical intervention, and subclinical control. Clinical participants are those who meet diagnostic criteria for one or more anxiety disorders, whereas subclinical participants present high self-reported anxiety but no mental disorder diagnosis. Intervention effects will based on self-report assessments conducted at pre-intervention, post-intervention (9 weeks later), and at 3-month follow-up.

This research will provide evidence regarding the suitability and effectiveness of TOUCHminds in promoting help-seeking among adolescents experiencing different levels of anxiety symptoms. Findings will contribute to the field of empirically validated web-based interventions tailored specifically for adolescents.

DETAILED DESCRIPTION:
Nearly 14% of adolescents experience mental health disorders, many of which remain unrecognized and untreated. Anxiety disorders, affecting approximately 5.5% of adolescents aged 15-19, commonly emerge during childhood or adolescence and are linked to anxiety persisting into adulthood, increased risk of other disorders such as substance abuse and major depressive disorder, and significant impairments across life domains, including reduced quality of life and lower educational attainment. Despite these risks, adolescents often show reluctance to seek help, particularly when symptoms are more severe. Barriers to help-seeking include lack of mental health literacy, which prevents from recognizing the severity of one's condition or from identifying it as a mental health issue, and mental health stigma, leading adolescents to conceal their struggles. Interventions often overlook additional barriers such as shame and low self-confidence. Promising facilitators for overcoming these barriers include fostering self-compassion, involving kindness and understanding towards oneself in difficult situations, and promoting well-being across emotional, psychological, and social dimensions. Additionally, enhancing readiness to change and utilizing motivational interviewing techniques, based on the transtheoretical model stages of change, may further facilitate adolescents' engagement in help-seeking behaviors by increasing motivation and managing ambivalence.

Interventions aimed at promoting adolescent help-seeking have typically been universal, potentially limiting their effectiveness for adolescents with clinical or subclinical symptoms who require more targeted support to recognize their need for professional help. Selective and indicated interventions, specifically tailored to these adolescents, have shown greater long-term efficacy but remain underexplored. Most existing programs primarily address barriers such as stigma and mental health literacy. Web-based interventions, particularly those that are multicomponent (e.g., psychoeducation, quizzes, vignettes) and involve minimal professional contact, have been suggested as effective in overcoming barriers such as stigma and low mental health literacy. However, key facilitators such as self-compassion, readiness for change and motivational interviewing techniques are largely absent from existing interventions, even though web-based interventions targeting self-compassion or integrating motivational interviewing appear to enhance their well-being and adolescents' engagement with mental health care.

TOUCHminds targets these gaps through a multicomponent web-based intervention, combined with synchronous psychologist-led sessions, addressing both help-seeking intentions and behaviors. The investigators will also assess changes in post-intervention and during follow-up, as the stability of change has been rarely explored in previous works targeting help-seeking. Additionally, the investigators aim to include adolescents with subclinical symptoms, often overlooked in existing programs. Finally, mechanisms of change remain unclear, particularly whether reduced stigma or improved mental health literacy drive help-seeking. Study I (feasibility) will assess recruitment procedures, dropout rates, usage patterns, therapist fidelity, acceptability, usability, satisfaction, and preliminary effects on help-seeking, in the precursors (mental health literacy, stigma, self-compassion, stage of change, readiness for change) of help-seeking and in well-being. Study II (RCT) will compare intervention groups (clinical, subclinical) with control groups across three moments. Expected results include increases in help-seeking intentions (both intervention groups), behaviors (intervention group clinical), precursors, and well-being, and changes in those precursors will explain shifts in intentions/behaviors over time.

All procedures will be authorized by the Directorate-General for Education, the General Data Protection Regulation of the University of Aveiro, and the University of Aveiro Ethics Committee for Clinical Research. Adolescents will be recruited in portuguese schools; adolescents and their guardians will receive full study information, confidentiality assurances, and will provide parental consent and adolescent assent, with no incentives. Screening comprises the State-Trait Anxiety Inventory for Children (STAIC) and a sociodemographic form; participants scoring 1 standard deviation above the mean will be invited to a Mini-KID diagnostic interview via videoconference to confirm inclusion/exclusion (i.e., include primary anxiety disorder and no diagnosis; exclude psychotic symptoms and suicidal risk). After completing the Mini-KID interview, the psychologist will complete the Clinical Global Impression - Severity scale (CGI-S) to provide a baseline assessment of psychopathology severity. Eligible participants will then be emailed to register to the platform, while adolescents outside criteria (e.g., psychotic symptoms, suicidal risk, other primary disorders) will be referred to school psychology services.

ELIGIBILITY:
Inclusion Criteria:

For all experimental and control groups, the inclusion criteria are:

* Aged between 15 and 17 years old at the time of screening;
* Fluent in Portuguese;
* Have access to a smartphone, tablet, or computer;
* Have reliable internet access.

Clinical Groups Specific:

* Must meet criteria for a primary diagnosis of at least one anxiety disorder, as assessed by the MINI-KID (Rijo et al., 2016).

Subclinical Groups Specific:

* Must not meet diagnostic criteria for any mental health disorder, as assessed by the MINI-KID (Rijo et al., 2016).

Exclusion Criteria:

Exclusion criteria for all experimental and all control groups are:

* Psychotic symptoms or suicidal risk as assessed via the Mini-Kid (Rijo et al., 2016);
* Being part of the special needs teaching system.
* Currently receiving psychological counselling.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2026-09-15 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
General Help-Seeking Questionnaire (GHSQ). | Administered one week before the intervention (T0), one week after completion (T1), and 3 months after completion (T2) in experimental groups (Studies I-II), and at corresponding times (9 weeks after T0 and 3 months later) in control groups (Study II).
  The GHSQ is a 12-item self-report scale that assesses adolescents' intentions to seek help for personal-emotional problems from various sources. Responses are rated on a 7-point Likert scale (1 = 'extremely unlikely' to 7 = 'extremely likely'). Its items refer to formal help (e.g., mental health professionals), semi-formal help (e.g., priests), informal help (e.g., partner), and self-help (e.g., the internet). sources. Higher scores indicate stronger intentions to seek help. The GHSQ has been adapted for use in Portugal and, despite the lack of formal psychometric studies, has been widely applied in research. For this study, the scale is further adapted to better reflect adolescents' social context. The adapted version includes formal help (e.g., psychologist), semi-formal help (e.g., teacher), informal help (e.g., friend), and self-help (e.g., online websites) sources. In addition, the original response option "I would not seek help from anyone" will be retaine.
Adolescent Help-Seeking Behavior Scale (AHSBS). | Administered one week before the intervention (T0), one week after completion (T1), and 3 months after completion (T2) in experimental groups (Studies I-II), and at corresponding times (9 weeks after T0 and 3 months later) in control groups (Study II).
  The AHSBS is a 17-item self-report scale developed for this study to assess how often adolescents seek help for emotional or psychological difficulties. Using the same items as the adapted GHSQ, but with new instructions, participants are asked to indicate how frequently they have turned to various sources of help in recent weeks. Responses are given on a 5-point Likert scale (1 = 'never' to 5 = 'always'). Help sources are categorized into formal, semi-formal, informal, and self-help. The total score reflects overall help-seeking frequency, with sub-scores available for each category. The AHSBS is currently under study for its psychometric properties and is expected to show good internal consistency, a structure consistent with help-seeking categories (formal, informal, semi-formal, and self-help), and construct validity in relation help-seeking intentions, stigma, and well-being.

SECONDARY OUTCOMES:
Adolescents' Mental Health Knowledge (AMHK). | Administered one week before the intervention (T0), one week after completion (T1), and 3 months after completion (T2) in experimental groups (Studies I-II), and at corresponding times (9 weeks after T0 and 3 months later) in control groups (Study II).
  The AMHK is a 15-item self-report scale assessing mental health literacy in adolescents, including symptom recognition, help-seeking, and attitudes toward mental health. Items (e.g., "If someone, over a period of time, avoids or misses school parties or oral presentations because they are afraid of being judged, to what extent do you consider it likely that they are experiencing symptoms of social anxiety?") are rated on a 4-point Likert-type scale ranging from 1 ("Very unlikely" or "Very useless") to 4 ("Very likely" or "Very useful"). It was adapted from the Mental Health Literacy Scale (MHLS) and developed with input from adolescents through think-aloud sessions to ensure developmental and cultural relevance. The measure is currently undergoing validation in a Portuguese adolescent sample to assess its internal consistency, construct validity, and factorial structure.
Peer Mental Health Stigmatization Scale (PMHSS). | Administered one week before the intervention (T0), one week after completion (T1), and 3 months after completion (T2) in experimental groups (Studies I-II), and at corresponding times (9 weeks after T0 and 3 months later) in control groups (Study II).
  The PMHSS is a 24-item self-report scale that assesses peer attitudes toward adolescents with mental health problems. Of these, 16 negative items measure two components: Stigma Agreement (personal endorsement of stigmatizing beliefs) and Stigma Awareness (perceptions of societal stigma). In this study, only these 16 items were used. Items (e.g., "Most people believe that young people with emotional or behavioral problems are dangerous") are rated on a 5-point Likert scale ranging from 'strongly disagree' to 'strongly agree'. Previous psychometric information indicates good internal consistency for the negative items and acceptable values for Stigma Agreement and Stigma Awareness. The Portuguese version is currently undergoing validation in an adolescent sample to assess its internal consistency, construct validity, and factorial structure.
Self-Compassion Scale for Adolescents (SCS-A). | Administered one week before the intervention (T0), one week after completion (T1), and 3 months after completion (T2) in experimental groups (Studies I-II), and at corresponding times (9 weeks after T0 and 3 months later) in control groups (Study II).
  The SCS-A is a 26-item self-report measure that assesses adolescents' self-compassion, defined as the ability to respond to personal difficulties with understanding and non-judgment. Items (e.g., "How I typically act toward myself in difficult times") are rated on a 5-point Likert scale (1 = 'almost never' to 5 = 'almost always'). The scale includes six subscales reflecting both compassionate (Self-Kindness, Common Humanity, Mindfulness) and uncompassionate (Self-Judgment, Isolation, Over-Identification) self-responding. Previous psychometric information on its Portuguese version indicates good internal consistency for the total scale and acceptable reliability for the subscales. Construct validity has been supported by positive associations with positive emotional memories and negative associations with symptoms of depression, anxiety, and stress.
University of Rhode Island Change Assessment (URICA). | Administered one week before the intervention (T0), one week after completion (T1), and 3 months after completion (T2) in experimental groups (Studies I-II), and at corresponding times (9 weeks after T0 and 3 months later) in control groups (Study II).
  The URICA is a 32-item self-report scale designed to evaluate motivation for behavior change across four stages: pre-contemplation, contemplation, action, and maintenance. Items (e.g., "I have been thinking that I could change something about myself") are rated on a 5-point Likert scale (1 = 'strongly disagree' to 5 = 'strongly agree'). Each stage is scored from 8 to 32, allowing identification of the individual's predominant stage. A readiness to change score is derived by summing the scores of contemplation, action, and maintenance, and subtracting the pre-contemplation score. Previous psychometric information indicates acceptable internal consistency for the total score in late adolescents and young adults, although subscale reliability was more variable. No analyses of item quality or factorial structure were previously performed. This measure is currently being further adapted and validated for use with Portuguese adolescents.
Mental Health Continuum - Short Form - for youth (MHC-SF). | Administered one week before the intervention (T0), one week after completion (T1), and 3 months after completion (T2) in experimental groups (Studies I-II), and at corresponding times (9 weeks after T0 and 3 months later) in control groups (Study II).
  The MHC-SF is a 14-item self-report scale for the assessment of adolescents' flourishing based on levels of subjective well-being: emotional, social, and psychological well-being. In response to the instruction ("Please answer the following questions about how you have been feeling during the past month"), participants rate each item (e.g., "How often do you felt happy?") using a 6-point Likert scale ranging from 0 = 'Never' to 5 = 'Every day'. Previous psychometric information indicates good internal consistency values and construct validity in relation to measures of quality of life, life satisfaction, anxiety, depression and internalizing and externalizing problems.

OTHER OUTCOMES:
Clinical Global Impression Scale (CGI). | Completed after the interview at baseline for all groups (CGI-S), and after each intervention session for experimental groups only (CGI-S and CGI-I; Studies I-II).
  The CGI is a clinician-rated measure designed to evaluate both the global severity of illness and changes in clinical status over time. It consists of three subscales: Severity of Illness (CGI-S), Global Improvement (CGI-I), and Efficacy Index. In the present study, only the CGI-S and CGI-I will be used. The CGI-S, which evaluates the severity of psychopathology, is rated on a seven-point scale, ranging from 1 = 'normal' to 7 = 'among the most extremely ill'. The CGI-I, which assesses the perceived change since the initiation of the intervention, is also rated on a seven-point scale, ranging from 1 = 'very much improved' to 7 = 'very much worse', and reflects clinical change relative to the participant's initial evaluation. For the current study, items were translated and adapted to European Portuguese by experts in clinical assessment and intervention, ensuring both linguistic and cultural adequacy.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Monteiro, M.Sc., Principal Investigator — William James Center for Research, Department of Education and Psychology, University of Aveiro.
Locations (1):
- William James Center for Research, Department of Education and Psychology, University of Aveiro., Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. (2024, October 10). Mental health of adolescents. https://www.who.int/news-room/fact-sheets/detail/adolescent-mental-health
- [Background] Woodward LJ, Fergusson DM. Life course outcomes of young people with anxiety disorders in adolescence. J Am Acad Child Adolesc Psychiatry. 2001 Sep;40(9):1086-93. doi: 10.1097/00004583-200109000-00018. PMID 11556633
- [Background] Wilson, C. J., Deane, F. P., Ciarrochi, J., & Rickwood, D. (2005). Measuring help-seeking intentions: Properties of the General Help-Seeking Questionnaire. Canadian Journal of Counselling, 39(1), 15-28.
- [Background] Werner-Seidler A, Perry Y, Calear AL, Newby JM, Christensen H. School-based depression and anxiety prevention programs for young people: A systematic review and meta-analysis. Clin Psychol Rev. 2017 Feb;51:30-47. doi: 10.1016/j.cpr.2016.10.005. Epub 2016 Oct 24. PMID 27821267
- [Background] van Doorn M, Nijhuis LA, Egeler MD, Daams JG, Popma A, van Amelsvoort T, McEnery C, Gleeson JF, Ory FG, Avis KA, Ruigt E, Jaspers MWM, Alvarez-Jimenez M, Nieman DH. Online Indicated Preventive Mental Health Interventions for Youth: A Scoping Review. Front Psychiatry. 2021 Apr 29;12:580843. doi: 10.3389/fpsyt.2021.580843. eCollection 2021. PMID 33995136
- [Background] Tuijnman A, Kleinjan M, Olthof M, Hoogendoorn E, Granic I, Engels RC. A Game-Based School Program for Mental Health Literacy and Stigma on Depression (Moving Stories): Cluster Randomized Controlled Trial. JMIR Ment Health. 2022 Aug 17;9(8):e26615. doi: 10.2196/26615. PMID 35976200
- [Background] Strawn JR, Lu L, Peris TS, Levine A, Walkup JT. Research Review: Pediatric anxiety disorders - what have we learnt in the last 10 years? J Child Psychol Psychiatry. 2021 Feb;62(2):114-139. doi: 10.1111/jcpp.13262. Epub 2020 Jun 5. PMID 32500537
- [Background] Schlack R, Peerenboom N, Neuperdt L, Junker S, Beyer AK. The effects of mental health problems in childhood and adolescence in young adults: Results of the KiGGS cohort. J Health Monit. 2021 Dec 8;6(4):3-19. doi: 10.25646/8863. eCollection 2021 Dec. PMID 35146318
- [Background] Sawyer MG, Borojevic N, Ettridge KA, Spence SH, Sheffield J, Lynch J. Do help-seeking intentions during early adolescence vary for adolescents experiencing different levels of depressive symptoms? J Adolesc Health. 2012 Mar;50(3):236-42. doi: 10.1016/j.jadohealth.2011.06.009. PMID 22325128
- [Background] Rijo D, Brazao N, Barroso R, da Silva DR, Vagos P, Vieira A, Lavado A, Macedo AM. Mental health problems in male young offenders in custodial versus community based-programs: implications for juvenile justice interventions. Child Adolesc Psychiatry Ment Health. 2016 Nov 1;10:40. doi: 10.1186/s13034-016-0131-6. eCollection 2016. PMID 27822300
- [Background] Prochaska, J. O., & DiClemente, C. C. (1982). Transtheoretical therapy: Toward a more integrative model of change. Psychotherapy: Theory, Research & Practice, 19(3), 276-288. https://doi.org/10.1037/h0088437
- [Background] Neto, D. D., Rocha, I., Figueiras, M. J., & Nunes Da Silva, A. (2021). Measuring Mental Health Literacy: Adaptation and Validation of the Portuguese Version of the Mental Health Literacy Scale (MHLS). European Journal of Mental Health, 16(1), 64-77. https://doi.org/10.5708/EJMH.16.2021.1.5
- [Background] Neff, K. (2003). Self-Compassion: An Alternative Conceptualization of a Healthy Attitude Toward Oneself. Self and Identity, 2(2), 85-101. https://doi.org/10.1080/15298860309032
- [Background] Miller, W. R., & Rollnick, S. (2013). Motivational interviewing: Helping people change (3rd ed.). Guilford Press.
- [Background] McKeague L, Hennessy E, O'Driscoll C, Heary C. Peer Mental Health Stigmatization Scale: psychometric properties of a questionnaire for children and adolescents. Child Adolesc Ment Health. 2015 Sep;20(3):163-170. doi: 10.1111/camh.12088. Epub 2015 Feb 16. PMID 32680400
- [Background] Matos, A. P., André, R. S., Cherpe, S., Rodrigues, D., Figueira, C., & Pinto, A. M. (2010). Estudo Psicométrico preliminar da Mental Health Continuum - Short Form - for youth numa amostra de adolescentes portugueses. Psychologica, 53, 131-156. https://doi.org/10.14195/1647-8606_53_7
- [Background] Martin A, Calhoun A, Paez J, Amsalem D. Destigmatizing perceptions about Black adolescent depression: randomized controlled trial of brief social contact-based video interventions. J Child Psychol Psychiatry. 2022 Nov;63(11):1270-1278. doi: 10.1111/jcpp.13570. Epub 2022 Jan 23. PMID 35066880
- [Background] Lemos, L. (2011). Motivação para a mudança de comportamentos de saúde [Dissertação de mestrado, Universidade de Aveiro]. Departamento de Educação, Universidade de Aveiro.
- [Background] Kutcher S, Wei Y, Coniglio C. Mental Health Literacy: Past, Present, and Future. Can J Psychiatry. 2016 Mar;61(3):154-8. doi: 10.1177/0706743715616609. No abstract available. PMID 27254090
- [Background] Krieger T, Martig DS, van den Brink E, Berger T. Working on self-compassion online: A proof of concept and feasibility study. Internet Interv. 2016 Oct 8;6:64-70. doi: 10.1016/j.invent.2016.10.001. eCollection 2016 Nov. PMID 30135815
- [Background] Keyes CL. The mental health continuum: from languishing to flourishing in life. J Health Soc Behav. 2002 Jun;43(2):207-22. PMID 12096700
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Kessler RC, Amminger GP, Aguilar-Gaxiola S, Alonso J, Lee S, Ustun TB. Age of onset of mental disorders: a review of recent literature. Curr Opin Psychiatry. 2007 Jul;20(4):359-64. doi: 10.1097/YCO.0b013e32816ebc8c. PMID 17551351
- [Background] Johnson JA, Devdutt J, Mehrotra S, Bhola P, Sudhir P, Sharma A. Barriers to Professional Help-seeking for Distress and Potential Utility of a Mental Health App Components: Stakeholder Perspectives. Cureus. 2020 Feb 28;12(2):e7128. doi: 10.7759/cureus.7128. PMID 32257673
- [Background] Howard KA, Griffiths KM, McKetin R, Ma J. Can a brief biologically-based psychoeducational intervention reduce stigma and increase help-seeking intentions for depression in young people? A randomised controlled trial. J Child Adolesc Ment Health. 2018 May;30(1):27-39. doi: 10.2989/17280583.2018.1467323. Epub 2018 May 15. PMID 29764293
- [Background] Horowitz JL, Garber J. The prevention of depressive symptoms in children and adolescents: A meta-analytic review. J Consult Clin Psychol. 2006 Jun;74(3):401-15. doi: 10.1037/0022-006X.74.3.401. PMID 16822098
- [Background] Hassett, A., & Isbister, C. (2017). Young men's experiences of accessing and receiving help from child and adolescent mental health services following self-harm. SAGE Open, 7(4), 1-10. https://doi.org/10.1177/2158244017745112
- [Background] Hassen HM, Behera MR, Jena PK, Dewey RS, Disassa GA. Effectiveness and Implementation Outcome Measures of Mental Health Curriculum Intervention Using Social Media to Improve the Mental Health Literacy of Adolescents. J Multidiscip Healthc. 2022 May 3;15:979-997. doi: 10.2147/JMDH.S361212. eCollection 2022. PMID 35535244
- [Background] Guy, W. (1976). ECDEU assessment manual for psychopharmacology (Publication No. ADM 76-338). U.S. Department of Health, Education, and Welfare, Public Health Service, Alcohol, Drug Abuse, and Mental Health Administration.
- [Background] Gulliver A, Griffiths KM, Christensen H, Brewer JL. A systematic review of help-seeking interventions for depression, anxiety and general psychological distress. BMC Psychiatry. 2012 Jul 16;12:81. doi: 10.1186/1471-244X-12-81. PMID 22799879
- [Background] Gulliver A, Griffiths KM, Christensen H. Perceived barriers and facilitators to mental health help-seeking in young people: a systematic review. BMC Psychiatry. 2010 Dec 30;10:113. doi: 10.1186/1471-244X-10-113. PMID 21192795
- [Background] Griffiths KM. Towards a framework for increasing help-seeking for social anxiety disorder. Aust N Z J Psychiatry. 2013 Oct;47(10):899-903. doi: 10.1177/0004867413493335. Epub 2013 Jun 6. No abstract available. PMID 23744983
- [Background] Gould MS, Greenberg T, Munfakh JL, Kleinman M, Lubell K. Teenagers' attitudes about seeking help from telephone crisis services (hotlines). Suicide Life Threat Behav. 2006 Dec;36(6):601-13. doi: 10.1521/suli.2006.36.6.601. PMID 17250466
- [Background] Fortune S, Sinclair J, Hawton K. Help-seeking before and after episodes of self-harm: a descriptive study in school pupils in England. BMC Public Health. 2008 Oct 24;8:369. doi: 10.1186/1471-2458-8-369. PMID 18947435
- [Background] Fonseca A, Moura-Ramos M, Canavarro MC. Attachment and Mental Help-Seeking in the Perinatal Period: The Role of Stigma. Community Ment Health J. 2018 Jan;54(1):92-101. doi: 10.1007/s10597-017-0138-3. Epub 2017 Apr 27. PMID 28451843
- [Background] Finlay-Jones AL, Parkinson A, Sirois F, Perry Y, Boyes M, Rees CS. Web-Based Self-Compassion Training to Improve the Well-Being of Youth With Chronic Medical Conditions: Randomized Controlled Trial. J Med Internet Res. 2023 Sep 13;25:e44016. doi: 10.2196/44016. PMID 37703081
- [Background] Figueiredo, D. V., Alves, F., & Vagos, P. (2024). Portuguese adapted version of the Clinical Global Impression Scale. [Unpublished manuscript].
- [Background] Essau CA, Lewinsohn PM, Olaya B, Seeley JR. Anxiety disorders in adolescents and psychosocial outcomes at age 30. J Affect Disord. 2014 Jul;163:125-32. doi: 10.1016/j.jad.2013.12.033. Epub 2014 Jan 2. PMID 24456837
- [Background] Essau CA, Lewinsohn PM, Lim JX, Ho MR, Rohde P. Incidence, recurrence and comorbidity of anxiety disorders in four major developmental stages. J Affect Disord. 2018 Mar 1;228:248-253. doi: 10.1016/j.jad.2017.12.014. Epub 2017 Dec 8. PMID 29304469
- [Background] Divin, N., Harper, P., Curran, E., Corry, D., & Leavey, G. (2018). Help-seeking measures and their use in adolescents: A systematic review. Adolescent Research Review, 3(1), 1-17. https://doi.org/10.1007/s40894-017-0078-8
- [Background] DiClemente CC, Schlundt D, Gemmell L. Readiness and stages of change in addiction treatment. Am J Addict. 2004 Mar-Apr;13(2):103-19. doi: 10.1080/10550490490435777. PMID 15204662
- [Background] Dias, P., & Gonçalves, M. (1999). Avaliação da ansiedade e da depressão em crianças e adolescentes (STAIC C2, CMAS-R, FSSC-R e CDI): Estudo normativo para a população portuguesa. In A. P. Soares, S. Araújo, & S. Caires (Eds.), Avaliação Psicológica: Formas e contextos (Vol. 6, pp. 553-564). Associação de Psicólogos Portugueses.
- [Background] Dean S, Britt E, Bell E, Stanley J, Collings S. Motivational interviewing to enhance adolescent mental health treatment engagement: a randomized clinical trial. Psychol Med. 2016 Jul;46(9):1961-9. doi: 10.1017/S0033291716000568. PMID 27045520
- [Background] Cunha, M., Xavier, A., & Castilho, P. (2016). Understanding self-compassion in adolescents: Validation study of the Self-Compassion Scale. Personality and Individual Differences, 93, 56-62. https://doi.org/10.1016/j.paid.2015.09.023
- [Background] Copeland WE, Angold A, Shanahan L, Costello EJ. Longitudinal patterns of anxiety from childhood to adulthood: the Great Smoky Mountains Study. J Am Acad Child Adolesc Psychiatry. 2014 Jan;53(1):21-33. doi: 10.1016/j.jaac.2013.09.017. Epub 2013 Oct 12. PMID 24342383
- [Background] Chandra A, Minkovitz CS. Stigma starts early: gender differences in teen willingness to use mental health services. J Adolesc Health. 2006 Jun;38(6):754.e1-8. doi: 10.1016/j.jadohealth.2005.08.011. PMID 16730608
- [Background] Bharadwaj, P., Pai, M. M., & Suziedelyte, A. (2017). Mental health stigma. Economics Letters, 159, 57-60. https://doi.org/10.1016/j.econlet.2017.06.028
- [Background] Andersson G, Titov N. Advantages and limitations of Internet-based interventions for common mental disorders. World Psychiatry. 2014 Feb;13(1):4-11. doi: 10.1002/wps.20083. PMID 24497236
- [Background] Amsalem D, Martin A. Reducing depression-related stigma and increasing treatment seeking among adolescents: randomized controlled trial of a brief video intervention. J Child Psychol Psychiatry. 2022 Feb;63(2):210-217. doi: 10.1111/jcpp.13427. Epub 2021 Apr 6. PMID 33821507
- [Background] Aguirre Velasco A, Cruz ISS, Billings J, Jimenez M, Rowe S. What are the barriers, facilitators and interventions targeting help-seeking behaviours for common mental health problems in adolescents? A systematic review. BMC Psychiatry. 2020 Jun 11;20(1):293. doi: 10.1186/s12888-020-02659-0. PMID 32527236